CLINICAL TRIAL: NCT01531192
Title: Zekai Tahir Burak Maternity Teaching Hospital, Ankara/Turkey
Brief Title: Comparison of Lactobacillus Reuteri and Nystatin Prophylaxis on Candida Colonization and Infection in Very Low Birth Weight Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Yekta, Principal Investigator, Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZTB630301
Record Dates: First submitted 2012-02-04; First posted 2012-02-10 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2012-02

CONDITIONS: Very Low Birth Weight Infants
Keywords: Lactobacillus reuteri; Nystatin; Very Low Birth Weight Infants; Candida Colonization
MeSH Terms: interventions — Nystatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactobacillus reuteri (Experimental): Lactobacillus reuteri 100 million CFU/day for 3 months
  Interventions: Dietary Supplement: Lactobacillus reuteri
- Nystatin (Active Comparator): 50000 unit/3 times a day
  Interventions: Drug: Nystatin

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri — Lactobacillus reuteri 100 million CFU/day for 3 months
  Other Names: BioGaia
  Arms: Lactobacillus reuteri
Drug: Nystatin — 50000 unit/3 times a day, both for orally and by orogastric route
  Other Names: Mikostatin
  Arms: Nystatin

SUMMARY:
Probiotics are favorable microorganisms that regulate the flora of the gastrointestinal system and stimulate the immune system. Lactobacillus reuteri was shown to reduce candida colonization. The objective of this study is to evaluate the efficacy of prophylactic Lactobacillus reuteri in reducing the candida colonization and infection in very low birth weight infants.

ELIGIBILITY:
Inclusion Criteria:

* Very low birth weight infants < 1500 gr
* Gestational age < 32 weeks

Exclusion Criteria:

* Genetic anomalies
* Short bowel syndrome
* Not willing to participate
* Allergy to Lactobacillus reuteri components

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Comparison of prophylactic Lactobacillus reuteri and nystatin on candida colonization and infection in very low birth weight infants | up to 6 months
  Rectal and skin swabs for Candida colonization will be taken weekly. Blood culture for Candida infection will be taken weekly.

SECONDARY OUTCOMES:
Effect of Lactobacillus reuteri on feeding intolerance | up to 6 months
  Feeding intolerance (gastric residuals in the amount that was more than half of the previous feeding, abdominal distention or heme-positive stools)
Effect of Lactobacillus reuteri on sepsis | up to 6 months
  Patients with culture positivity will accept as proven sepsis.
Effect of Lactobacillus reuteri on length of hospital stay | up to 6 months
  Specified length of hospital stay as days.
Effect of Lactobacillus reuteri on necrotizing enterocolitis in VLBW infants | up to 6 months
  NEC diagnosis will make modified Bell's criteria. Grade 1A will not include in NEC group.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Yekta Oncel, MD, Principal Investigator — Neonatology
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Division of Neonatology, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Oncel MY, Arayici S, Sari FN, Simsek GK, Yurttutan S, Erdeve O, Saygan S, Uras N, Oguz SS, Dilmen U. Comparison of Lactobacillus reuteri and nystatin prophylaxis on Candida colonization and infection in very low birth weight infants. J Matern Fetal Neonatal Med. 2015;28(15):1790-4. doi: 10.3109/14767058.2014.968842. Epub 2014 Oct 9. PMID 25245226
- See also: Lactobacillus reuteri — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=L040030000&QV1=LACTOBACILLUS+REUTERI
- See also: Nystatin — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0001400619&QV1=NYSTATIN